CLINICAL TRIAL: NCT01826903
Title: Perinatal Depression Treatment and Child Development: A Follow-Up of the Thinking Healthy Programme
Brief Title: Perinatal Depression Treatment and Child Development
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Human Development Research Foundation, Pakistan (Other); Grand Challenges Canada (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00034166; Saving Brains #0058 (Other Grant/Funding Number: Grand Challenges Canada); ISRCTN65316374 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2013-03-26; First posted 2013-04-09 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Depression
Keywords: Depression; Cognitive Behavior Therapy; Child Development
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- depressed mother/child dyad - intervention
- depressed mother/child dyad - no intervention
- non-depressed mother/child dyad

SUMMARY:
The purpose of this study is to examine whether the successful perinatal depression intervention among mothers (Thinking Healthy Programme, THP) has led to improved developmental outcomes in the children 6 years later. Economic and human resources aspects of the intervention will also be evaluated to determine overall societal benefits from investment in such a program, feasibility of scaling up the intervention and its sustainability in the long-term. The primary hypothesis is that children of mothers who participated in the THP will have better cognitive outcomes and socio-emotional functioning when compared to children of mothers randomized to the control group.

ELIGIBILITY:
Inclusion Criteria:

* children of women who were eligible to participate in the Thinking Healthy Programme

Exclusion Criteria:

* developmental disability, visual or hearing impairment

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes children of women who participated in the Thinking Healthy Programme and children of women who were eligible for participation in the Thinking Healthy Programme but who screened negative for depression at the time.
Sampling Method: Probability Sample
Enrollment: 964 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Estimate of general intelligence | Re-enrollment visit, approximately 7 years post-intervention
Measures of executive functions | Re-enrollment visit, approximately 7 years post-intervention
  Working memory, cognitive flexibility, inhibitory control, and sustained attention will be measured by standard tests of cognitive functioning.
Level of literacy and numeracy | Re-enrollment visit, approximately 7 years post-intervention
Presence of behavioral and emotional problems (socio-emotional development) | Re-enrollment visit, approximately 7 years post-intervention

SECONDARY OUTCOMES:
Height-for-age | Re-enrollment visit, approximately 7 years post-intervention
Weight-for-age | Re-enrollment visit, approximately 7 years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Maselko, ScD, Principal Investigator — Duke University; Siham Sikander, PhD, Principal Investigator — Human Development Research Foundation, Pakistan
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

REFERENCES:
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313